CLINICAL TRIAL: NCT01958034
Title: Bilberry as a Dietary Supplement After Myocardial Infarction (The BEAR SMART Trial)
Acronym: BEAR SMART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Ole Frobert, MD, PhD, MD, PhD, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-06-05
Record Dates: First submitted 2013-09-27; First posted 2013-10-08 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Vaccinium myrtillus extract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary supplement with bilberry extract (Experimental): Billberry powder 3 times daily for 2 months.
  Interventions: Dietary Supplement: Bilberry extract
- Control (No Intervention): No dietary supplement with bilberry extract

INTERVENTIONS:
Dietary Supplement: Bilberry extract
  Arms: Dietary supplement with bilberry extract

SUMMARY:
In a double blinded, randomized, clinical trial of patients suffering from STEMI (ST-segment elevation myocardial infarction) or non-STEMI (non-ST-segment elevation myocardial infarction)compare the effect of 3 months of dietary supplement with bilberry extract on a range of parameters with prognostic importance in cardiovascular disease: lipids, inflammation, oxidative stress and heart function.

Following inclusion of 8 individuals and as of February 12, 2014: Due to intolerance to "bilberry placebo powder" we have amended to the protocoll that the trial design is changed from blinded to open and that the bilberry arm of the trial carries on in an open design and that the control group will receive no dietary supplement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of STEMI as defined by chest pain suggestive for myocardial ischemia for at least 30 minutes before hospital admission, time from onset of symptoms of less than 24 hours, and an ECG with new ST-segment elevation in two or more contiguous leads of ≥0.2 mV in leads V2-V3 and/or ≥0.1 mV in other leads or a probable new-onset left bundle branch block.
* Patients with a diagnosis of non-STEMI as defined by a combination of; onset of symptoms such as central chest pain or an aggravated angina pectoris, with or without an ECG change with ST-segment lowering or an inverted T-wave, and at least two values with levels of troponin-T or troponin-I above the established margin of an MI.

Exclusion Criteria:

* Need for emergency coronary artery bypass grafting
* Inability to provide informed consent
* Age below 18 years
* Previous randomization in the BEAR SMART trial
* A daily intake, or the intent to start a daily intake of bilberries in some form (fresh berries, bilberry powder, bilberrysoup etc)

Exclusion Criteria:

* Need for emergency coronary artery bypass grafting
* Inability to provide informed consent
* Age below 18 years
* Previous randomization in the BEAR SMART trial
* A daily intake, or the intent to start a daily intake of bilberries in some form (fresh berries, bilberry powder, bilberrysoup etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
6 minutes walk test | 2 months
  The effect of intervention on a standardized physical challenge - the 6 minutes walk test

SECONDARY OUTCOMES:
C-reactive protein | Baseline and 2 months
  The effect of intervention on the inflammatory marker CRPö
Inflammatory markers and markers of heart function | Baseline and 2 months
  The effect of intervention on markers of inflammation: IL-6 (interleukin 6), TNF-α (tumor necrosis factor α), INF-γ (interferon γ), markers of oxidative stress: oxidized LDL, carbonylated proteins, 2-OHDG, H2O2, hexanoyl L lysine, nitrogen oxide synthase (NOS), markers of myocardial damage and heart failure: BNP (brain natriuretic peptide) and troponin I, markers of endothelial function: VEGF (vascular endothelial growth factor), 8-isoprostane, E-selectin, measures of plasma lipids; total cholesterol, LDL-cholesterol, TGA (triacylglycerides), and measures of patient compliance and biological effect of bilberry supplementation: quercetin,

CONTACTS AND LOCATIONS:
Overall Officials: Ole Frobert, MD, PhD, Principal Investigator — Department of Cardiology, Orebro University Hospital, Sweden
Locations (1):
- Department of Cardiology, Orebro University Hospital, Örebro, Örebro County, Sweden

REFERENCES:
- [Derived] Arevstrom L, Bergh C, Landberg R, Wu H, Rodriguez-Mateos A, Waldenborg M, Magnuson A, Blanc S, Frobert O. Freeze-dried bilberry (Vaccinium myrtillus) dietary supplement improves walking distance and lipids after myocardial infarction: an open-label randomized clinical trial. Nutr Res. 2019 Feb;62:13-22. doi: 10.1016/j.nutres.2018.11.008. Epub 2018 Nov 17. PMID 30803503